CLINICAL TRIAL: NCT04836403
Title: Validation of the Chinese Version of the Sinus and Nasal Quality of Life Survey (SN-5) and Correlation With Pediatric Obstructive Sleep Apnea and Asthma
Brief Title: Validation of the Chinese Version of the Sinus and Nasal Quality of Life Survey (SN-5)
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH105-REC1-138(AR-1)
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Chronic Rhinosinusitis
Keywords: SN-5; Quality of life; children

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rhinosinusitis without treatment group: children aged 2 and 12 years with rhinosinusitis not receiving treatment
  Interventions: Other: Sinus and nasal quality of life survey questionnaire (SN-5)
- Rhinosinusitis with treatment group: children aged 2 and 12 years with rhinosinusitis receiving treatment
  Interventions: Other: Sinus and nasal quality of life survey questionnaire (SN-5)
- healthy volunteers: children aged 2 and 12 years without rhinosinusitis
  Interventions: Other: Sinus and nasal quality of life survey questionnaire (SN-5)

INTERVENTIONS:
Other: Sinus and nasal quality of life survey questionnaire (SN-5) — The SN-5 consists of five questions on a 7-point scale that assesses the frequency of the following symptoms: (1) nasal obstruction, (2) sinus infection, (3) allergies, (4) emotional distress, and (5) activity limitations. The scoring system is as follows: 1 indicates "none of the time," 2 indicating "hardly any time at all," 3 indicates "a small part of the time," 4 indicates "some of the time," 5 indicates "a good part of the time," 6 indicates "most of the time," and 7 indicates "all of the time." Higher scores indicate more severe sinonasal symptoms. One item from a global faces scale scored from 0 to 10 is used to evaluate overall QoL related to nasal or sinus disease. Higher scores on this scale indicate a less severe impact of nasal or sinus disease. The scores from the first five items (1-7 each)

SUMMARY:
The purpose of our study was to validate the Chinese version of the Sinus and Nasal Quality of Life Survey (SN-5)and correlation with the incidence of pediatric obstructive sleep apnea and asthma.

The study will enroll pediatric patients of rhino-sinusitis and their parents to finish Questionnaire 1, including Chinese version of SN-5, visual analogue scale (VAS), Pediatric allergy disease Pediatric Allergic Disease Quality of Life Questionnaire (PADQLQ), OSA-18 quality of Life Survey, and asthma-diagnostic questionnaire . Some patients re-tested SN-5 in 1 week later. After four weeks, participants finish these questionnaire 2, including SN-5, VAS, and PADQLQ. In addition, the author will invite health children without rhino-sinusitis disease and their parents to fill in Questionnaire 1. The Chinese version of SN-5 will be validated to establish its reliability and validity.

DETAILED DESCRIPTION:
The purpose of the study was to validate the Chinese version of the Sinus and Nasal Quality of Life Survey (SN-5)and correlation with the incidence of pediatric obstructive sleep apnea and asthma.

The study will enroll pediatric patients of rhino-sinusitis and parents to finish Questionnaire 1, including Chinese version of SN-5, visual analogue scale (VAS), Pediatric allergy disease Pediatric Allergic Disease Quality of Life Questionnaire (PADQLQ), OSA-18 quality of Life Survey, and asthma-diagnostic questionnaire . Some patients re-tested SN-5 in 1 week later. After four weeks, they finish these questionnaire 2, including SN-5, VAS, and PADQLQ. In addition, the author will invite health children without rhino-sinusitis disease and their parents to fill in Questionnaire 1. The Chinese version of SN-5 will be validated to establish its reliability and validity.

From December 2016 to December 2017, healthy volunteers and children with persistent sinonasal symptoms were enrolled. Guardians of the participants completed the SN-5, a visual analog scale (VAS) of nasal symptoms, and the Obstructive Sleep Apnea-18 (OSA-18) ; the responses were used to assess internal consistency, discriminant validity, and treatment responsiveness. A nontreatment group was administered the SN-5 1 week later to assess test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

Children with one or more of the following symptoms, purulent nasal discharge, nasal congestion, cough, or postnasal drip for at least 1 month.

Exclusion Criteria:

* craniofacial anomalies
* cognitive deficits
* illiteracy in traditional Chinese.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Rhinosinusitis patients were recruited from pediatric clinics practicing Western or Chinese medicine
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Test-retest reliability | 1 week
  A nontreatment group was administered the SN-5 1 week later to assess test-retest reliability.
Concurrent validity | baseline
  The correlation between SN-5 and VAS scores was used to analyze the concurrent validity of the SN-5.
Discriminant validity | baseline
  Discriminant validity was assessed by calculating the difference between the SN-5 scores for participants with rhinosinusitis and for the healthy participants. These differences were analyzed with the Mann-Whitney U test.

SECONDARY OUTCOMES:
the mean scores of SN-5 | 4 week
  To evaluate the responsiveness of the treatment , the author compare the mean score of treatment group after 4-week-treatment compared to baseline mean score of SN-5 before treatment.Data analyzed with the Wilcoxon signed-rank test. Effects were evaluated through intention-to-treat analysis.
correlation with score of SN-5 and score of OSA-18 quality of life questionnaire (OSA-18) | baseline and 4 week
  To evaluate the correlation of SN-5 and OSA-18, Spearman correlation coefficients between the SN-5 and OSA-18 scores were analyzed.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lai WY, Kay DJ, Wei CC, Huang FW, Liang KL, Yen HR. Validation of the traditional Chinese version of the Sinus and Nasal Quality of Life Survey (SN-5) for children. Pediatr Neonatol. 2022 Jul;63(4):410-417. doi: 10.1016/j.pedneo.2022.01.008. Epub 2022 May 2. PMID 35595617